CLINICAL TRIAL: NCT01101477
Title: Target-Controlled Infusion of Propofol for Flexible Bronchoscopy Sedation: Determining the Optimal Titrating Regimen
Brief Title: Target-Controlled Infusion of Propofol for Flexible Bronchoscopy Sedation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Hypoxemia(SPaO2<80%) episodes occured significantly in the arm titration by 0.5ug/ml
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, 林定佑, Attending physician, Lecture of Medicine, Division of Thoracic Medicine, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 98-3441A3
Record Dates: First submitted 2010-04-07; First posted 2010-04-12 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-11

CONDITIONS: Flexible Bronchoscopy
Keywords: Target-controlled infusion,; bronchoscopy,; sedation,; propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Titration by target effect site concentration (Cet) 0.5μg/ml (Active Comparator): The investigator will titrate the Cet to keep stable vital signs and sedative level during the flexible bronchoscopy. The criteria for titration is descried in the intervention.
  Interventions: Procedure: TCI titration by different Cet.
- Titration by Cet 0.2μg/ml (Active Comparator): The investigator will titrate the Cet to keep stable vital signs and sedative level during the flexible bronchoscopy. The criteria for titration is descried in the intervention.
  Interventions: Procedure: TCI titration by different Cet.
- Titration by Cet 0.1μg/ml (Active Comparator): The investigator will titrate the Cet to keep stable vital signs and sedative level during the flexible bronchoscopy. The criteria for titration is descried in the intervention.
  Interventions: Procedure: TCI titration by different Cet.

INTERVENTIONS:
Procedure: TCI titration by different Cet. — Induction:
  After topical xylocaine and alfentanil 5μg/kg iv 1 minute before, Cet 2.0μg/ml is started on the TCI pump ('Vial" Injectomat TIVA Agilia syringe infusion pump, Fresenius Kabi, France). The sedative level will be accessed by sedation scale "OAA/S" every 30 seconds till OAA/S ≦3(Responds only to name called loudly). The current Ce will be set as the maintenance Cet.
  If desired OAA/S is not achieved after reaching 2.0μg/ml,Cet will be increased every 90 seconds by the regimens be assigned until OAA/S ≦3. The current Ce will be set as the maintenance Cet.
  Maintenance:
  The Cet will be increased according to the assigned regimens if:
  1. Patients become irritant and interfere procedures.
  2. Patients open eyes or talk to express uncomfortable.
  The Cet will be decreased if:
  1. Systolic blood pressure is less than 90mmHg;
  2. Mean arterial blood pressure is less than 65mmHg;
  3. Oxyhemoglobin saturation is less than 90 %
  with any duration.

SUMMARY:
Flexible bronchoscopy (FB) sedation requires keeping sedative level in a narrow window to prevent over or under sedation. Sedative drug titration according to subjective adjustment by individual physician may cause unsteady drug concentration. Target controlled infusion (TCI) has been provided a precise pharmacokinetic control of propofol, direct control the effect side, (eg. Brain) concentration (Ce), and been applied in surgical anesthesia and variable procedure sedation. We designed this pilot study to evaluate the optimal regimen of TCI in FB sedation.

DETAILED DESCRIPTION:
Propofol is ideal for bronchoscopy sedation because of its fast onset and quick recovery effect. Our research and reports from different investigators demonstrate that patients received propofol sedation recover fast with excellent satisfaction for bronchoscopy. However, the amount of propofol for induction and maintenance is calculated simply by patient's body weight and physicians' experience. For those non-anesthesiologists, who perform sedative work outside the operating room, and inexperienced anesthesiologist without fully considering the individual pharmacokinetic and pharmacodynamic differences may generate unstable drug plasma concentration and increase cardio-respiration suppression. Therefore, a manner which can assess and measure objectively individual pharmacokinetic differences may improve the sedative quality and decrease the complication rate.

A model called "Target-controlled infusion"(TCI), built from massive pharmacokinetic samples of propofol, could now give precise pharmacokinetic control. Several pharmacokinetic models built-in in TCI, includes the Schnider model which use concentration of effect site (Ce, the propofol concentration in the brain) as the sedative guide. The model integrates individual variants of age, height, weight and gender to calculate the infusion profile to achieve predetermined steady "target effect site concentration" (Cet). Because of the unique consideration of individual pharmacokinetic variants and Ce targeting, TCI provides predictable sedative level and is suitable for procedures requiring narrowing therapeutic level. Beside general anesthesia, TCI has been applied in breast biopsy, upper gastrointestinal endoscopic ultrasound and endoscopic retrograde cholangiopancreatography at outpatient clinic. According to these evidences, there is potential role of TCI in bronchoscopic sedation.

Based on current evidence and our experience, we design this study to evaluate the optimal regimen for induction and procedure during bronchoscopy. We hope this study could provide the more safety and efficient bronchoscopic sedation for patients and physicians.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years old or more) required elective flexible bronchoscopy and sedation.

Exclusion Criteria:

* American Society of Anesthesiologists classification of physical status 4 and 5, including hepatic or renal failure, severe obstructive sleep apnea and severe chronic obstructive pulmonary disease.
* Mallampati score 4 or 5.
* Significant Central nervous system disorders or other factors contributing to access consciousness difficultly.
* Men with body mass index(BMI) large than 42，Females with BMI large than 35.
* Allergic history to study drugs.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Yu Lin, MD, Principal Investigator — Department of Thoracic Medicine, Chang Gung Memorial hospital
Locations (1):
- Department of Thoracic Medicine, Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Background] Fanti L, Agostoni M, Arcidiacono PG, Albertin A, Strini G, Carrara S, Guslandi M, Torri G, Testoni PA. Target-controlled infusion during monitored anesthesia care in patients undergoing EUS: propofol alone versus midazolam plus propofol. A prospective double-blind randomised controlled trial. Dig Liver Dis. 2007 Jan;39(1):81-6. doi: 10.1016/j.dld.2006.09.004. Epub 2006 Oct 16. PMID 17049322
- [Derived] Lin TY, Lo YL, Hsieh CH, Ni YL, Wang TY, Lin HC, Wang CH, Yu CT, Kuo HP. The potential regimen of target-controlled infusion of propofol in flexible bronchoscopy sedation: a randomized controlled trial. PLoS One. 2013 Apr 24;8(4):e62744. doi: 10.1371/journal.pone.0062744. Print 2013. PMID 23638141

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing elective flexible bronchoscopy (FB) and sedation were screened for enrolment at the bronchoscopic room on the day of exam.
Pre-assignment Details: If patients or accompanying family refused to paticipate anytime before assignment to groups.
Period: Overall Study
Arm/Group | Titration by Target Effect Site Concentration (Cet) 0.5μg/ml | Titration by Cet 0.2μg/ml | Titration by Cet 0.1μg/ml
Started | 49 | 49 | 46
Completed | 44 | 46 | 45
Not Completed | 5 | 3 | 1
Not completed — Protocol Violation | 5 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Titration by Target Effect Site Concentration (Cet) 0.5μg/ml | Titration by Cet 0.2μg/ml | Titration by Cet 0.1μg/ml | Total
Number analyzed (Participants) | 49 | 49 | 46 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 28 | 21 | 76
  >=65 years | 22 | 21 | 25 | 68
Age Continuous [Mean (Standard Deviation); unit: years] | 61.4 (13.0) | 62.6 (13.5) | 63.4 (14.4) | 62.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 22 | 67
  Male | 26 | 27 | 24 | 77
Region of Enrollment [Number; unit: participants]
  Taiwan | 49 | 49 | 46 | 144

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Hypoxemia During Flexible Bronchoscopy
Description: Hypoxemia is defined as:
  Oxyhemoglobin saturation (SPO2) is less than 90 % with any duration
Time Frame: During sedative induction and bronchoscopy
Population: The participants who received intervention completely were analyzed.
Measure: Number; unit: participants
Arm/Group | Titration by Target Effect Site Concentration (Cet) 0.5μg/ml | Titration by Cet 0.2μg/ml | Titration by Cet 0.1μg/ml
Number analyzed (Participants) | 44 | 46 | 45
participants | 29 | 22 | 18
Statistical Analysis 1: Comparison: Titration by Target Effect Site Concentration (Cet) 0.5μg/ml vs Titration by Cet 0.2μg/ml vs Titration by Cet 0.1μg/ml; The patients with at lease one episode of hypoxemia (SPaO2<90%) during FB were analyzed by Chi-square test. P value less 0.05 means significance, 2-sided; Test type: Superiority or Other; p = 0.05, Chi-squared

2. Primary Outcome: The Number of Changes in Target Effect Site Concentration During Flexible Bronchoscopy
Description: The investigator will titrate the target effect site concentration (Cet) during bronchoscopy according to protocol to keep stable vital signs and sedative levels. The numbers of adjustment will be recorded to show which regimen required less adjustment to keep stable sedative levels and vital signs.
Time Frame: During sedative induction and bronchoscopy
Reporting Status: Not Posted

3. Secondary Outcome: The Recovery Time to Orientation
Description: The recovery time to orientation was defined as the time between finishing bronchoscopy to the time when the patients could spontaneously open their eyes, recall their date of birth, and correctly perform finger-nose test.
Time Frame: after bronchosocpy
Reporting Status: Not Posted

4. Secondary Outcome: The Total Doses of Propofol During Induction and Overall Procedures
Description: The dosses of propofol used during induction and overall flexible bronchoscopy will be recored from the screen of the TCI pump.
Time Frame: after bronchoscopy
Reporting Status: Not Posted

5. Secondary Outcome: The Cooperation of Patients From the View of Bronchoscopists
Description: After the bronchoscopy, the bronchoscopist will be asked by 10-point Verbal Analogus Scale (0: the best cooperation, 10: the worst cooperation) to express how they fell about the cooperation of patients undergoing the bronchoscopy.
Time Frame: After bronchoscopy
Reporting Status: Not Posted

6. Secondary Outcome: The Global Tolerance for Flexible Bronchoscopy
Description: After the recovery, patients will be asked about the tolerance of bronchoscopy performed to them by 10-point Verbal Analogus Scale (0: best tolerance, 10: worst tolerance)
Time Frame: After recovery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the starting of induction to patients leaving the bronchoscopic room after recovery.
Arm/Group | Titration by Target Effect Site Concentration (Cet) 0.5μg/ml | Titration by Cet 0.2μg/ml | Titration by Cet 0.1μg/ml
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/46 | 0/45
Other Adverse Events (participants affected / at risk) | 6/44 | 1/46 | 2/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Titration by Target Effect Site Concentration (Cet) 0.5μg/ml (N=44) | Titration by Cet 0.2μg/ml (N=46) | Titration by Cet 0.1μg/ml (N=45)
oxyhemoglobin saturation (SpO2) less than 80% (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 2

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No